CLINICAL TRIAL: NCT04741737
Title: Repeat Sentinel Lymph Node Biopsy in Ipsilateral Breast Tumor Recurrence Without Distant Metastasis: A Single-arm, Multicenter, Prospective Study
Brief Title: Repeat Sentinel Lymph Node Biopsy in Ipsilateral Breast Tumor Recurrence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2020-0448
Record Dates: First submitted 2021-01-28; First posted 2021-02-05 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Mastectomy
Keywords: Breast cancer, Recurrence, Sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- reSLNB arm (Experimental): repeat SLNB procedure is performed in when the patient is diagnosed with ipsilateral breast tumor recurrence, who had undergone partial mastectomy and sentinel lymph node biopsy for primary operation.
  Interventions: Procedure: reSLNB arm

INTERVENTIONS:
Procedure: reSLNB arm — Radioisotope, blue dye, dual mapping methods are all allowed for re-SLNB mapping. Positive finding in re-SLNB is defined according to AJCC 8th edition, as micrometastasis or macrometastasis. Isolated tumor cell is considered negative. When sentinel lymph node is not identified, axillary operation is via physician's choice. When re-SLNB finding is negative, no further axillary lymph node dissection is performed. If there is node metastasis from re-SLNB, axillary lymph node dissection or radiation therapy can be performed as in physician's choice.

SUMMARY:
According to the standard treatment guidelines established until recently, in the case of ipsilateral breast tumor recurrence without systemic metastasis, salvage mastectomy or lumpectomy can be performed when either partial or whole breast radiation therapy is possible. On the other hand, there are currently no standard treatment guidelines for axillary treatment, and the evidence for this is limited. Axillary lymph node metastasis was reported to occur in about 26% of breast cancer patients who had negative sentinel lymph nodes from previous surgery for primary breast cancer and only local recurrence occurred. It is still important in the decision of treatment or adjuvant radiation therapy. However, it is known that most of the patients with ipsilateral breast recurrence do not have axillary lymph node metastasis. Therefore, performing axillary axillary surgery in all of these patients does not help the patient's survival in many cases, but rather can lead to complications such as lymphedema and seroma and postoperative wound infection. A question about the implementation of axillary lymph node resection has been raised and for this reason, it is necessary to study whether surveillance lymph node biopsy is still effective in patients with recurrence in the ipsilateral breast.

Most of the studies on ipsilateral breast tumor recurrence without systemic metastasis reported to date are case reports or small retrospective studies. In addition, the combined meta-analysis also has limitations in that the study design is not uniform, and there are many cases in which primary breast cancer surgery performed total mastectomy or axillary lymph node dissection. This study is a multicenter prospective study designed to validate the clinical effectiveness of repeat-SLNB conducted in patients with ipsilateral breast tumor recurrence among patients who previously underwent breast conservation and sentinel lymph node biopsy for unilateral primary breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 19 years old
2. Patients who are expected to undergo surgery under the diagnosis of ipsilateral breast tumor recurrence(histologically confirmed in situ disease or invasive disease)
3. Patients who had partial mastectomy and sentinel lymph node biopsy for prior operation for the initially diagnosed breast cancer
4. Patients considered to be axillary lymph node negative from clinical findings
5. Patients who understand and willingly participate in the study

Exclusion Criteria:

1. Patients with recurrence in other regions. (e.g. ipsilateral axillary lymph node, supraclavicular lymph node, internal mammary lymph node, etc.)
2. Patients who are not eligible to perform SLNB
3. Patients who received mastectomy or axillary lymph node dissection for prior operation
4. Patients who experienced recurrence within a year from the primary operation
5. Patientes who are known to have axillary lymph node metastasis before the secondary operation, histologically confirmed from tissue biopsy or cytology
6. Patients with systemic recurrence
7. Patients with inflammatory breast cancer

5) Pregnant and lactating patients

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
5 year disease free survival | 5 years after surgery (re-SLNB)
  To prove non-inferiority of re-SLNB compared to ALND regarding disease free survival

SECONDARY OUTCOMES:
identification rate of sentinel lymph node | 5 years after surgery
  identification rate of sentinel lymph node
5-year overall survival | 5 years after surgery
  5-year overall survival
5-year local recurrence free survival | 5 years after surgery
  5-year local recurrence free survival
5-year regional recurrence free survival | 5 years after surgery
  5-year regional recurrence free survival
5-year distant metastasis free survival | 5 years after surgery
  5-year distant metastasis free survival
survival by adjuvant treatment | 5 years after surgery
  survival analysis according to the adjuvant treatment after secondary surgery
survival by tumor subtype | 5 years after surgery
  survival analysis by tumor subtype
identification rate of sentinel lymph node by tumor location | 5 years after surgery
  identification rate of sentinel lymph node according to the location of primary tumor(caudal/non-caudal)
5-year DFS by tumor location | 5 years after surgery
  5-year DFS accoridng to the location of primary tumor (caudal/non-caudal)

CONTACTS AND LOCATIONS:
Overall Officials: Joon Jeong, Principal Investigator — Gangnam Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea